CLINICAL TRIAL: NCT06318312
Title: Effects of Different Hypoxia Exposures on Cognitive Performance in Healthy Adults
Brief Title: Effects of Hypoxia on Cognitive Performance
Acronym: HYPCOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HYP_MR_2024
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Hypoxia
Keywords: cognitive; anticipation; memory; attention; reaction time
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 11% FiO2 (Experimental): Hypoxic exposure: fraction of oxygen inspired (FiO2) = 11% (~5100 m, ~16735 ft)
  Interventions: Other: Hypoxia
- 13% FiO2 (Experimental): Hypoxic exposure: fraction of oxygen inspired (FiO2) = 13% (~3800 m, ~12470 ft)
  Interventions: Other: Hypoxia
- 15% FiO2 (Experimental): Hypoxic exposure: fraction of oxygen inspired (FiO2) = 15% (~2750 m, ~9000 ft)
  Interventions: Other: Hypoxia
- PLA / 21% FiO2 (Placebo Comparator): Hypoxic exposure / placebo condition: fraction of oxygen inspired (FiO2) = 21% (sea level)
  Interventions: Other: Hypoxia

INTERVENTIONS:
Other: Hypoxia — Hypoxic exposure: FiO2 = 11% Hypoxic exposure: FiO2 = 13% Hypoxic exposure: FiO2 = 15% Hypoxic exposure / placebo: FiO2 = 21%
  Other Names: hypoxic exposure

SUMMARY:
The goal of this clinical trial is to determine the effects of different hypoxia exposures (FiO2 = 11%, 13%, 15%, and 21%) on cognitive performance in healthy adults. The main questions it aims to answer are:

* What is the best hypoxia exposure to improve reaction time, anticipation, attention and memory tasks?
* Which hypoxia exposure causes the greatest detriments in cognitive function?

DETAILED DESCRIPTION:
Participants will completed four trials in a single-blinded crossover randomised control trial. In the first session, individuals familiarised with the different cognitive tests and hypoxic exposures. In the next four experimental trials (separated by 1 week), participants arrived at the laboratory and rested in a seated for 10 min. The vital signs (i.e., SpO2, HR, blood pressure) and Lake Louise Score were recorded prior to mask placed and start with in one of the four conditions: a) PLA/NOR, b) FiO2=15%, c) FiO2=13% or FiO2=11%. In this hypoxic condition the participant will spend a total of 45 min, of which 30 min was at rest, and the other 15 min was performing the cognitive tasks (i.e., memory test, go/no-go test, eriksen flanker test, anticipation task and reaction time test).

ELIGIBILITY:
Inclusion Criteria:

* Physically active individuals ( >150 min/week moderate physical activity or >75 min/week vigorous physical activity)
* Non-smokers
* Individuals without serious and undiagnosed health problems

Exclusion Criteria:

* Pregnancy and/or breastfeeding
* Residing at an altitude of more than 1300 m
* Having been exposed to an altitude of more than 900 m in the last 8 months
* Having performed a study with hypoxia in the last 8 months
* Suffering from any of the following diseases/pathologies: diabetes, sleep apnoea, dyslexia, colour blindness, blurred vision, respiratory and/or neuromuscular diseases.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Memory | During each hypoxic condition
  To study the modulation of memory storage processes, three 20-item word lists were created. Each word in the list will be presented for 5 s. This will be followed by a 100 s memory consolidation interval, after which there will be a 120 s period in which as many words as the participants can remember will be written down (First time). After 15 min, participants will perform a recall task (Second time) in which they will have to rewrite all the words they remember at that time.
Attention | During each hypoxic condition
  The ability of maintaining the attention and inhibiting an appropriate response will be measured by "Go/No-Go Test" [fastest, slowest, and average response time (in seconds), and successful attempts (percentage; %)] and "Eriksen Flanker Test" [congruent and incongruent reaction time (in seconds)].
Anticipation | During each hypoxic condition
  Visual acuity related to hand-eye coordination and anticipation will be assessed using the Bassin Anticipation Timer instrument. The best anticipation time (in seconds) of each condition (5, 10 and 15 mph) will be taken.
Reaction time | During each hypoxic condition
  Reaction time (in seconds) shall be assessed with the Dynavision™ D2 Visomotor Device using the "Reaction Time Test". In this test the fastest visual, motor and physical reaction time will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Performance and Sport Rehabilitation Laobratory. University of Castilla-La Mancha, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No